CLINICAL TRIAL: NCT00582530
Title: Serum Protein Profiling to Characterize Patient Risk in Men Undergoing Radical Prostatectomy
Brief Title: Men Undergoing Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 04-132
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Early Prostate Cancer; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood

GROUPS / COHORTS (1):
- 1 men with prostate cancer: Patients who have opted for radical prostatectomy as treatment for prostate cancer.
  Interventions: Other: Whole Blood Draw

INTERVENTIONS:
Other: Whole Blood Draw — The plan is to obtain the research blood sample at the time of routine preoperative and postoperative blood testing, typically performed 1-2 weeks prior to surgery and then again 6 weeks to 12 months after surgery

SUMMARY:
The purpose of this study is to see if the protein pattern in your blood can predict whether or not your prostate tumor is aggressive. We will use a new and very sensitive technique, called mass spectroscopy, to measure hundreds of pieces of protein in your blood. A computer will make a picture of the protein pattern. We will do this in 500 men before their prostate surgery and see if there is a pattern that predicts what the tumor looks like under the microscope. We will also check the protein pattern in your blood 6 weeks to 12 months after the surgery to see if your pattern changes.

DETAILED DESCRIPTION:
In this pilot study, we propose to address the question: is there a small peptide mass proteomic profile/pattern in blood that can distinguish men with a clinically insignificant/latent prostate cancer from men with more advanced pathological features? We will obtain a pre-operative blood sample from men with clinically localized prostate cancer undergoing radical prostatectomy and determine their preoperative small peptide mass proteomic profile. The pathological features of the radical prostatectomy will be determined and the patient will be classified as having either a pathologically insignificant/latent prostate cancer or a significant cancer. We will then analyze whether or not the small peptide mass proteomic profile in blood can distinguish these groups before radical prostatectomy. In addition, each of these patients will have a blood sample collected at least 6 weeks to 12 months after surgery to evaluate and compare changes that occur as a result of radical prostatectomy. This will determine the effect of radical prostatectomy on the small peptide mass proteomic profile in blood and determine if the proteomic profiles in blood collected prior to radical prostatectomy can identify men at increased risk for recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older with clinically localized prostate cancer (cT1- T2NxM0)
* Scheduled for radical prostatectomy
* Prostate biopsy at least 6 weeks prior to scheduled radical prostatectomy
* Signed, informed consent
* Patient must be able to attend both the preoperative and postoperative blood draws.

Exclusion Criteria:

* A period of less than 6 months prior/current treatment with hormonal therapy (LHRH agonist/antagonist, antiandrogen, 5-alpha-reductase inhibitor).
* A period of less than 6 months prior/current treatment with an alpha-blocker

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology Clinic at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2004-12-28 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
To determine if men with pathologically latent prostate cancer have a different preoperative proteomic profile than men with a pathologically significant cancer. | conclusion of study

SECONDARY OUTCOMES:
To determine the effect of radical prostatectomy on the proteomic profile in blood samples from men with a pathologically latent cancer. This should suggest the contribution of 'benign'prostate to the small peptide proteomic profile in blood. | conclusion of study
To determine the effect of radical prostatectomy on the protein profile in blood samples from men with pathologically significant cancer. This should (in combination with 2) suggest the contribution of prostate cancer to the proteome in blood samples. | preoperative and postoperative
Determine if pre-tx small peptide proteomic profile in blood collected prior to rad. prostatectomy can ident men at increased risk for recurrence, compared to only using the postop nomogram to assess risk of biochem recur after radical prostatectomy | preoperative and postoperative
Determine the impact of sample type on proteomic results, will obtain both coagulated & anti-coagulated samples & perform these studies in parallel to examine which collect method might prove the optimal source for improving our predictive models. | preoperative and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org